CLINICAL TRIAL: NCT01081665
Title: A Two-year, Post-marketing Observational Study to Follow-up Patients With End Stage Renal Disease Undergoing Haemodialysis, Receiving Zemplar for Prevention and Treatment of Secondary Hyperparathyroidism
Brief Title: Follow-up Patients With End Stage Renal Disease Receiving Zemplar to Prevent and Treat Secondary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P06-120
Record Dates: First submitted 2010-02-27; First posted 2010-03-05 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Kidney Failure; Secondary Hyperparathyroidism
Keywords: Chronic Kidney Failure; Secondary Hyperparathyroidism; Paricalcitol IV treatment; Safety and efficacy assessment
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Kidney Disease: All eligible patients treated with IV Paricalcitol (Zemplar)

SUMMARY:
The aim of this post-marketing observational study is to obtain further data on the long term use, safety and efficacy of Zemplar as it is prescribed in the normal clinical setting and according to the approved Summary of Product Characteristics for the treatment of secondary hyperparathyroidism in hemodialysis patients in Greece.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety of Zemplar® in the treatment of Secondary hyperparathyroidism (iParathormone>300 pg/mL) in subjects on hemodialysis treated in conditions of usual clinical care.

The primary safety endpoints of this study are to evaluate the safety of Zemplar by recording the number of hospitalizations and days hospitalized.

A secondary efficacy endpoint will be the proportion of subjects achieving therapeutic success. Therapeutic success with Zemplar® will be defined as:

* 40% reduction in the base iPTH level is achieved, and/or;
* serum iParathormone level < 300 pg/mL.

Additional secondary endpoints are the incidence (proportion of patients) of clinically meaningful hypercalcemia (defined as corrected serum calcium (Ca) > 11.0 mg/dL taken at 2 consecutive measurements), hyperphosphatemia (defined as serum phosphorous (P)>6.5 mg/dL taken at 2 consecutive measurements), and elevated Ca x P product (defined as serum Ca x P>65 mg^2/dL^2 taken at 2 consecutive measurements). Safety also will be assessed through adverse event monitoring and evaluation of laboratory variables and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >= 18 years of age and diagnosed with secondary hyperparathyroidism and a pretreatment iParathormone > 300 pg/mL.
* Subject is receiving chronic hemodialysis.
* Subject for which treatment with Zemplar Injection is indicated clinically according to the criteria of participating investigator.
* Subject has provided their informed consent to participate.

Exclusion Criteria:

* Subject has a corrected serum calcium > 10.5 mg/dL, serum phosphorus >= 6.5 mg/dL or subjects with corrected Ca x P >= 65 mg^2/dl^2.
* Subject has known hypersensitivity and/or toxicity to vitamin D metabolites and/or other product ingredients.
* Subject has participated in clinical study within the last month.
* Zemplar is contraindicated according to the Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with secondary hyperparathyoidism treated with IV Paricalcitol according to the approved Summary of Product Characteristics
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2006-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Xynos, MD, Study Chair — Abbott Laboratories Hellas S.A.
Locations (19):
- Greece (19):
  - Site Reference ID/Investigator# 32055, Athens
  - Site Reference ID/Investigator# 32050, Athens
  - Site Reference ID/Investigator# 32051, Athens
  - Site Reference ID/Investigator# 32049, Athens
  - Site Reference ID/Investigator# 5283, Athens
  - Site Reference ID/Investigator# 32056, Chalcis
  - Site Reference ID/Investigator# 32057, Chania
  - Site Reference ID/Investigator# 32077, Cholargós
  - Site Reference ID/Investigator# 32058, Drama
  - Site Reference ID/Investigator# 32076, Katerini
  - Site Reference ID/Investigator# 32059, Kavala
  - Site Reference ID/Investigator# 32053, Komotini
  - Site Reference ID/Investigator# 32060, Lamia
  - Site Reference ID/Investigator# 32061, Lefkada
  - Site Reference ID/Investigator# 32062, Livadia
  - Site Reference ID/Investigator# 32048, Piraeus
  - Site Reference ID/Investigator# 32054, Preveza
  - Site Reference ID/Investigator# 32063, Ptolemaida
  - Site Reference ID/Investigator# 32075, Volos

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Kidney Disease
Started | 237
Full Analysis Set | 237
Evaluable Population | 212 (Participants with baseline and at least 2 post-baseline parathormone measurements at 24 months.)
Completed | 142
Not Completed | 95
Not completed — Death | 41
Not completed — Lost to Follow-up | 18
Not completed — Withdrawal by Subject | 17
Not completed — Change of dialysis unit | 10
Not completed — Regulation of iPTH | 5
Not completed — Change in renal replacement therapy | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 237
Age Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 127
Region of Enrollment [Number; unit: participants]
  Greece | 237
Age at chronic kidney disease diagnosis [Mean (Standard Deviation); unit: years] — The age of participants when they were diagnosed with chronic kidney disease. Based on data reported by 222 participants.
  years | 53.6 (14.7)
Time since chronic kidney disease diagnosis [Mean (Standard Deviation); unit: years] — The amount of time elapsed from the time the participant was diagnosed with chronic kidney disease to study entry. Based on data reported by 222 participants.
  years | 8.8 (6.8)
Time since starting haemodialysis [Mean (Standard Deviation); unit: years] — At study entry, the amount of time that had elapsed from participants first starting haemodialysis, a procedure that filters the blood to remove harmful wastes.
  years | 3.6 (4.4)
Time since diagnosis of secondary hyperparathyroidism [Mean (Standard Deviation); unit: years] — At study entry, the amount of time that had elapsed since participants were first diagnosed with hyperparathyroidism, a condition where the parathyroid glands make too much parathyroid hormone, causing an imbalance of calcium and phosphorous in the body. Based on data reported by 228 participants.
  years | 2.0 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation of Paricalcitol by Recording the Number of Hospitalizations
Description: The number of participants who were hospitalized during the study and the number of hospitalizations are summarized.
Time Frame: Baseline to Month 24 Visit
Population: Analysis included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 237
participants
  Participants with no hospitalizations | 152
  Participants with at least 1 hospitalization | 85
  >Participants with 1 hospitalization | 59
  >Participants with 2 hospitalizations | 16
  >Participants with 3 or more hospitalizations | 10

2. Secondary Outcome: The Proportion of Patients Achieving Therapeutic Success (Defined as 40% Reduction in Base Parathormone Level and/or Parathormone Level <300 pg/ml)
Description: Therapeutic success of paricalcitol treatment was defined as a 40% decrease from the baseline measurement in the level of intact parathyroid hormone (also known as iPTH or parathormone) and/or a serum intact parathyroid hormone level less than 300 picograms per milliliter (pg/mL) for at least 2 consecutive available measurements during the 24-month follow-up period.
Time Frame: Baseline to Month 24 Visit
Population: Analysis based on the evaluable population, defined as participants with baseline and at least 2 post-baseline parathormone measurements at the 24-month post-treatment follow-up visit.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 212
percentage of participants | 78.3

3. Secondary Outcome: The Incidence of Clinically Significant Hypercalcemia
Description: The number of participants with clinically significant hypercalcemia (too much calcium in the blood), defined as a corrected serum calcium level greater than 11.0 milligrams per deciliter (mg/dL) at 2 consecutive measurements.
Time Frame: Baseline to Month 24 Visit
Population: Analysis included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 237
Participants | 16

4. Secondary Outcome: The Incidence of Clinically Significant Hyperphosphatemia
Description: The number of participants with clinically significant hyperphosphatemia (too much phosphorous in the blood), defined as serum phosphorous levels greater than 6.5 milligrams per deciliter (mg/dL) at 2 consecutive measurements.
Time Frame: Baseline to Month 24 Visit
Population: Analysis included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 237
Participants | 107

5. Secondary Outcome: The Incidence of Clinically Significant Elevation of Calcium-phosphorous (Ca x P) Product
Description: The number of participants with clinically significant levels of calcium-phosphorous product (Ca x P), defined as serum calcium-phosphorous product levels greater than 65 milligrams squared per deciliters squared (mg^2/dL^2) at 2 consecutive measurements.
Time Frame: Baseline to Month 24 Visit
Population: Analysis included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 237
Participants | 81

6. Secondary Outcome: To Estimate the Incidence of (S)AEs/(S)ADRs
Description: The number of adverse events, serious adverse events (including death), adverse drug reactions, and serious adverse drug reactions experienced by participants during the study are summarized. Adverse events include any events reported regardless of whether or not they were considered related to the study drug. Adverse drug reactions include events where a causal relationship between the drug and the occurence of the event is suspected. For additional details see the Reported Adverse Events section.
Time Frame: Baseline to Month 24 Visit
Population: Analysis included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 237
participants
  Experienced an adverse event (serious/non-serious) | 196
  >Experienced non-serious adverse event | 170
  >Experienced serious adverse event | 94
  Experienced non-serious adverse drug reaction | 127
  Experienced serious adverse drug reaction | 10
  Total number of deaths reported | 43
  >Number of deaths during the study | 41
  >Number of deaths after study completion | 2
  Death considered related to study drug | 2

7. Primary Outcome: Safety Evaluation of Paricalcitol by Recording the Number of Days Hospitalized
Description: The mean (average) number of days hospitalized per participant for those hospitalized during the study.
Time Frame: Baseline to Month 24 Visit
Population: Based on participant hospitalizations during the study where the length of hospitalization was known (82 participants total).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 82
days | 16.1 (17.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected and reported from the time the participant signed the informed consent form until the end of the study. Participants were treated with Zemplar for an average of 19 months during the study.
Arm/Group | Chronic Kidney Disease
Serious Adverse Events (participants affected / at risk) | 94/237
Other Adverse Events (participants affected / at risk) | 170/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease (N=237)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 12
Acute myocardial infarction (Cardiac disorders) | 8
Cardio-respiratory arrest (Cardiac disorders) | 7
Angina pectoris (Cardiac disorders) | 5
Chest pain (Cardiac disorders) | 5
Atrial fibrillation (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Palatal oedema (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 15
Chills (General disorders) | 3
Death (General disorders) | 2
Medical device complication (General disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 1
Treatment failure (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Gallbladder oedema (Hepatobiliary disorders) | 1
Respiratory tract infection (Infections and infestations) | 10
Septic shock (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 2
Gangrene (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Enterobacter bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fistula (Injury, poisoning and procedural complications) | 1
Vascular access infection (Injury, poisoning and procedural complications) | 1
Blood calcium increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Hematocrit increased (Investigations) | 1
Weight decreased (Investigations) | 1
Fluid retention (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 3
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Femur fracture (Musculoskeletal and connective tissue disorders) | 1
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 1
Necrotising fasciitis (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalitis (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Intracranial haematoma (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Communication disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Renal cyst ruptured (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Haemorrhage (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Femoral artery occlusion (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Ischemia (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Poor venous access (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease (N=237)
Anaemia (Blood and lymphatic system disorders) | 9
Respiratory tract infection (Infections and infestations) | 6
Catheter site infection (Infections and infestations) | 3
Calcium phosphate product increased (Investigations) | 84
Blood phosphorous increased (Investigations) | 27
Haematocrit decreased (Investigations) | 14
Blood parathyroid hormone decreased (Investigations) | 9
Blood calcium increased (Investigations) | 8
Haematocrit increased (Investigations) | 6
Serum ferritin decreased (Investigations) | 5
Blood pressure increased (Investigations) | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 107
Hypercalcaemia (Metabolism and nutrition disorders) | 19
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Anxiety disorder (Psychiatric disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.